CLINICAL TRIAL: NCT02981238
Title: Descriptive Study of a Phytotherapy Strategy for Sleep Disorders Related to Anxiety With Phytostandard® Eschscholtzia and Valerian, a Dietary Supplement Based on Eschscholtzia and Valerian Extracts
Brief Title: Phytotherapy Strategy for Sleep Disorders Related to Anxiety With a Combination of Eschscholtzia and Valerian Extracts
Status: Completed | Type: Observational
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Other Study IDs: PiL-Obs-SLEE-PI-015
Record Dates: First submitted 2016-11-22; First posted 2016-12-05 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Sleep Disorders Related to Anxiety
MeSH Terms: interventions — Valeriana extract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Phytostandard® Eschscholtzia / Valerian

SUMMARY:
The aim of the study is to evaluate the effect of a one-month supplementation with Phytostandard® Eschscholtzia and valerian on the Insomnia Severity Index (ISI), in insomniac so-called adjustment subjects (occasional or short-term insomnia)

DETAILED DESCRIPTION:
For this study, 40 patients are going to be included. They will have a supplementation of Phytostandard® Eschscholtzia and valerian, from 2 to 4 tablets per day during 28 days.

on the one hand, during the two visits (inclusion and follow-up), the investigator completes the Hamilton Anxiety Scale (HAM-A). During the inclusion visit, he completes with his patient the epworth scale.

on the other hand, patients complete ISI twice : just after the inclusion visit and just before the follow-up visit. He completes two sleep schedules, the first one during the first week of complement and the second one during the fourth.

ELIGIBILITY:
Inclusion Criteria of patients:

* Currently having sleep disorders related to an anxiety and / or having some in the last 3 months
* Having an alteration of sleep on the previous month which results in a score strictly greater than 7 according to the index of Severity of Insomnia (ISI)
* For which the investigator freely advises his patient a complement with Phytostandard® Eschscholtzia and Valerian
* For which the patient freely agrees to complement itself after advice of his doctor with Phytostandard® Eschscholtzia and Valerian
* Having been informed of the study and accepting the collection and processing of their data

Exclusion Criteria:

* Suffering from an anxiety resulting in a HAM-A score (Hamilton Anxiety Rating Scale) greater than or equal to 30
* With a score on Epworth's sleepiness scale strictly greater than 10 (suggestive of a major hypersomnia)
* Presenting symptoms of sleep apnea syndrome
* Presenting symptoms of a restless legs syndrome
* Presenting a chronic pain syndrome requiring the daily intake of analgesic(s)
* Under psychotropic treatment (neuroleptic, anxiolytic, antidepressant or hypnotic) or under treatment to alter the waking state (antihistamines, beta-blockers, some cough syrups, etc.)

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from sleep disorders linked to anxiety
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
evolution of the Index of Severity of Insomnia (ISI) | day 0 and day 28
  This outcome is compared with ISI at day 0 : we compared both the global score and each item scores

SECONDARY OUTCOMES:
Evolution of Hamilton Anxiety Scale (HAM-A) | day 0 and day 28
  This outcome is compared with HAM-A at day 0
Percentage of Satisfaction | day 28
  using a likert scale of satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Pileje Network of general practitioners, Paris, France